CLINICAL TRIAL: NCT00806871
Title: Local Steroid Injection in the Treatment of Idiopathic Carpal Tunnel Syndrome: A Randomized Double-blind Placebo-controlled Trial Among Patients Planned for Surgical Treatment
Brief Title: Steroid Injection Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: prövningsprotokoll 080723
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2011-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Methylprednisolone; Methylprednisolone Acetate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: Methylprednisolone 40 mg
- B (Active Comparator)
  Interventions: Drug: Methylprednisolone 80 mg
- C (Placebo Comparator)
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Methylprednisolone 40 mg — Depo-medrol 40 mg , suspension, injection in the carpal tunnel, one time use
  1 ml 40 mg Methylprednisolone + 1 ml 10mg Lidocaine + 1 ml saline
  Other Names: Depo-medrol
  Arms: A
Drug: Methylprednisolone 80 mg — Depo-medrol 80 mg , suspension, injection in the carpal tunnel, one time use.
  2 ml 80mg Methylprednisolone + 1 ml 10mg Lidocaine
  Other Names: Depo-medrol
  Arms: B
Drug: Sodium chloride — Saline solution 0,9%, injection in the carpal tunnel, one time use
  1 ml 10 mg Lidocaine + 2 ml saline
  Other Names: Saline; NaCl
  Arms: C

SUMMARY:
The aim of this study is to assess the efficacy of injecting steroid into the carpal tunnel in relieving symptoms of carpal tunnel syndrome for at least 1 year with outcomes measured with patient evaluated symptoms score.Out of the patients referred by primary care, those with a clinical diagnosis of CTS who have tried wrist splint and whose symptom severity is judged by the examining surgeon to warrant surgery are offered to be put on the waiting list for carpal tunnel release. This means a waiting time of approximately 3 months. Patients who give informed consent will be asked to attend the outpatient clinic for a physical examination followed by allocation to one of the three trial groups. Immediately following the allocation the patients will receive the assigned treatment.

DETAILED DESCRIPTION:
www.biomedcentral.com/1471-2474/11/76

ELIGIBILITY:
Inclusion Criteria:

* Primary, idiopathic CTS
* Age 18-70 years, either gender
* Symptom duration of at least 3 months and inadequate response to wrist splint
* Symptoms of classic or probable CTS according to the diagnostic criteria in Katz hand diagram
* Nerve conduction studies showing median neuropathy at the wrist and no other abnormalities or, in the absence of abnormal nerve conduction study results, 2 surgeons should independently diagnose the patient with CTS.
* Scheduled for carpal tunnel release (ie, symptom severity indicating need for surgery)exclusion criteria

Exclusion Criteria:

* Previous steroid injection for CTS in the same wrist
* Inflammatory joint disease, diabetes mellitus· Vibration-induced neuropathy, polyneuropathy
* Pregnancy
* Trauma to the affected hand in the previous year
* Previous CTS surgery in the affected hand
* Inability to complete questionnaires due to language problem or cognitive disorder
* Severe medical illness
* Known abuse of drugs and/or alcohol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2008-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The CTS symptom severity score after treatment. | 10 weeks
Rate of surgery | 52 weeks

SECONDARY OUTCOMES:
The CTS symptom severity score after treatment | 52 weeks
Time to surgery | 52 weeks
QuickDASH score | 52 weeks
SF-6D score | 52 weeks
Patient satisfaction with the results of treatment (VAS scale) | 52 weeks
Registration of adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Isam Atroshi, MD, PhD, Study Chair — Lund university, department of clinical sciences, Hässleholm hospital, department of orthopedics
Locations (1):
- Ortopediska kliniken, sjukvårdsorganisationen Hässleholm/CSK, Hässleholm, Sweden

REFERENCES:
- [Background] Atroshi I, Gummesson C, Johnsson R, Ornstein E, Ranstam J, Rosen I. Prevalence of carpal tunnel syndrome in a general population. JAMA. 1999 Jul 14;282(2):153-8. doi: 10.1001/jama.282.2.153. PMID 10411196
- [Background] Atroshi I, Gummesson C, Johnsson R, McCabe SJ, Ornstein E. Severe carpal tunnel syndrome potentially needing surgical treatment in a general population. J Hand Surg Am. 2003 Jul;28(4):639-44. doi: 10.1016/s0363-5023(03)00148-5. PMID 12877853
- [Background] Wintman BI, Winters SC, Gelberman RH, Katz JN. Carpal tunnel release. Correlations with preoperative symptomatology. Clin Orthop Relat Res. 1996 May;(326):135-45. PMID 8620634
- [Background] Ahlberg J, Johansson H, Widenfalk B. [Disabling injuries following carpal tunnel syndrome surgery]. Lakartidningen. 2007 Oct 3-9;104(40):2884-6. No abstract available. Swedish. PMID 17966804
- [Background] Benson LS, Bare AA, Nagle DJ, Harder VS, Williams CS, Visotsky JL. Complications of endoscopic and open carpal tunnel release. Arthroscopy. 2006 Sep;22(9):919-24, 924.e1-2. doi: 10.1016/j.arthro.2006.05.008. PMID 16952718
- [Background] Marshall S, Tardif G, Ashworth N. Local corticosteroid injection for carpal tunnel syndrome. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD001554. doi: 10.1002/14651858.CD001554.pub2. PMID 17443508
- [Derived] Hofer M, Ranstam J, Atroshi I. Extended Follow-up of Local Steroid Injection for Carpal Tunnel Syndrome: A Randomized Clinical Trial. JAMA Netw Open. 2021 Oct 1;4(10):e2130753. doi: 10.1001/jamanetworkopen.2021.30753. PMID 34677593
- [Derived] Atroshi I, Flondell M, Hofer M, Ranstam J. Methylprednisolone injections for the carpal tunnel syndrome: a randomized, placebo-controlled trial. Ann Intern Med. 2013 Sep 3;159(5):309-17. doi: 10.7326/0003-4819-159-5-201309030-00004. PMID 24026316
- [Derived] Flondell M, Hofer M, Bjork J, Atroshi I. Local steroid injection for moderately severe idiopathic carpal tunnel syndrome: protocol of a randomized double-blind placebo-controlled trial (NCT 00806871). BMC Musculoskelet Disord. 2010 Apr 21;11:76. doi: 10.1186/1471-2474-11-76. PMID 20409331